CLINICAL TRIAL: NCT00006301
Title: Evaluation of the Immune Response in Humans After Exposure to Hepatitis C Virus
Brief Title: Immune Response to Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000221; 00-DK-0221
Record Dates: First submitted 2000-09-27; First posted 2000-09-28 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2015-03-24

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Viral Sequence; PCR; T Cell; Seroconversion; Cytokines
MeSH Terms: conditions — Hepatitis C; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will identify and characterize immune factors involved in hepatitis C infection and elimination of the virus. Individual responses to hepatitis C infection vary; some people are able to eliminate the virus, whereas others remain chronically infected. This study may identify factors important in preventing infection that may be of help in developing a vaccine or more effective treatments.

People over 18 years old who have been exposed to hepatitis C virus may participate in this study. Subjects will be recruited from the National Institutes of Health, Inova Fairfax Hospital, Occupational Medical Services-IDP P.C., Washington Hospital Center and Holy Cross Hospital, all in the Washington, D.C. metropolitan area. Individual patients from other centers will also be recruited on a case by case basis.

Participants will have 40 to 60 cc (1 to 2 ounces) of blood drawn at seven intervals. The first collection will be as soon as possible after exposure to hepatitis C virus and then again at 2, 4, 6, 12, 24, and 48 weeks after exposure. The white blood cells will be studied for their response to the virus, and markers for infection will be followed. If infection develops, additional samples of blood may be requested, and patients will be offered evaluation for treatment. Test results will be kept confidential and will not be entered into any medical records.

DETAILED DESCRIPTION:
The course and outcome of hepatitis C virus (HCV) infection is determined by both host and viral factors, none of which have been well defined. In this study, we will follow and assess patients who are occupationally exposed to HCV for viral and immunologic factors that may relate to disease outcome. This protocol is mostly a sample acquisition protocol to support laboratory research. Patients will be interviewed and have blood (and lymphocytes) taken as soon as possible after exposure and again after 2, 4, 6, 12, 24 and 48 weeks. Virological markers, serum antibodies and both CD4 and CD8 T cell responses to HCV will be monitored. Persons who develop hepatitis C will be referred for therapy or enrolled in therapeutic trials currently in place at the National Institutes of Health. These studies will help define the relative roles of virological and immunological factors in determining the course and outcome of HCV infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or female;

All ethnic groups;

Age above 18 years;

Defined exposure to hepatitis C.

EXCLUSION CRITERIA:

Subjects with a Hct of less than 30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2000-09-24; Study Completion 2015-03-24

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (5):
- United States (5):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Holy Cross Hospital, Silver Spring, Silver Spring, Maryland
  - Occupational Medicine Services, Annandale, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Background] Puro V, Petrosillo N, Ippolito G. Risk of hepatitis C seroconversion after occupational exposures in health care workers. Italian Study Group on Occupational Risk of HIV and Other Bloodborne Infections. Am J Infect Control. 1995 Oct;23(5):273-7. doi: 10.1016/0196-6553(95)90056-x. PMID 8585637
- [Background] Arai Y, Noda K, Enomoto N, Arai K, Yamada Y, Suzuki K, Yoshihara H. A prospective study of hepatitis C virus infection after needlestick accidents. Liver. 1996 Oct;16(5):331-4. doi: 10.1111/j.1600-0676.1996.tb00755.x. PMID 8938635
- [Background] Mizuno Y, Suzuki K, Mori M, Hayashi K, Owaki T, Hayashi H, Kumada K, Ohba K, Mizokami M. Study of needlestick accidents and hepatitis C virus infection in healthcare workers by molecular evolutionary analysis. J Hosp Infect. 1997 Feb;35(2):149-54. doi: 10.1016/s0195-6701(97)90103-1. PMID 9049819